CLINICAL TRIAL: NCT01166230
Title: An Open, Non-interventional, Retrospective, Comparative, Multicenter Follow-up Study in Patients Included in the Previously Completed Clinical Study PCB305/04, to Assess Longer-term Recurrence Rates in Patients After Hexvix® (Cysview®)Fluorescence Cystoscopy/Transurethral Resection of the Bladder (TURB) or White Light Cystoscopy/TURB
Brief Title: Longer-term Recurrence Rates in Patients With Bladder Cancer After Hexvix (Cysview)Fluorescence Cystoscopy/TURB
Status: Completed | Type: Observational
Sponsor: Photocure (Industry)
Responsible Party: Sponsor
Other Study IDs: PC B305/E10
Record Dates: First submitted 2010-07-19; First posted 2010-07-20 (Estimated); Results first posted 2013-11-14 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-03

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Ta/T1, randomized to white light cystoscopy: Patients with non-invasive papillary bladder cancer (Ta/T1), enrolled in the previously completed pivotal phase III study PC B305/04 who were followed for recurrence.
- Patients with Ta/T1 randomized to Hexvix cystoscopy: Patients with non-invasive papillary bladder cancer (Ta/T1), enrolled in the previously completed pivotal phase III study PC B305/04 who were followed for recurrence.

SUMMARY:
The study is intended to investigate whether the improved initial detection and resection of bladder cancer lesions in patients with non-muscle invasive bladder cancer with Hexvix (Cysview) fluorescence cystoscopy/TURB will lead to a longer-term reduction in recurrences compared to standard white light cystoscopy/TURB.

DETAILED DESCRIPTION:
A previously completed pivotal clinical study PC B305/04 demonstrated reduced recurrence rates for patients with papillary bladder cancer who underwent Hexvix (Cysview) and white light cystoscopy and transurethral resection (TURB) of the bladder compared to patients who underwent white light cystoscopy and TURB alone.

The present study is intended to investigate whether the improved initial detection and resection of bladder cancer lesions in patients with non-muscle invasive bladder cancer with Hexvix (Cysview) fluorescence cystoscopy/TURB will also lead to a longer-term reduction in recurrences compared to standard white light cystoscopy/TURB.

No safety data was collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients of study PC B305/04 with Ta or T1, that were followed for recurrence are eligible to be included in this study.

Exclusion Criteria:

* Patient died during clinical study PC B305/04

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-invasive papillary bladder cancer, enrolled in the previously completed pivotal phase III study PC B305/04, who were followed for recurrence will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 551 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Barton Grossman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (24):
- United States (14):
  - Stanford Cancer Center, Department of Urology, Stanford, California
  - V.A. Medical Center, Gainesville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - South Florida Clinical Research Center, Inc., Pembroke Pines, Florida
  - The Emory Clinic, Dept of Urology, Atlanta, Georgia
  - Boston University School of Medicine, Boston, Massachusetts
  - Urologic Clinical Research Unit, Gonda 7102, Mayo Clinic Rochester, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mount Sinai Medical Center, Department of Urology, New York, New York
  - URMC, Rochester, New York
  - Thomas Jefferson Medical College, Department of Neurology, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Department of Urologic Surgery, Nashville, Tennessee
  - Baylor College of Medicine, Scott Department of Urology, Houston, Texas
  - The University of Texas MD Anderson cancer center, Houston, Texas
- AKH, Klinik für Urologie der Universität Wien, Vienna, Austria
- Canada (2):
  - Kingston General Hospital, Kingston, Ontario
  - CHUQ Hotel-Dieu de Quebec, Québec
- Germany (5):
  - University Clinic of Giessen, Department of Urology, Giessen
  - Klinikum der Universität München-Großhardern, Urologische Klinik und Poliklinik, München
  - Urologische Klinik München-Planegg, Planegg
  - Akadem. Lehrkrankenhaus der Uni Regensburg, Klinik für Urologie, Regensburg
  - Universitätsklinik Tuebingen, Universitätsklinik für Urologie, Tübingen
- Netherlands (2):
  - Department of Urology, Academic Medical Center, University of Amsterdam, Amsterdam
  - Department of Urology, UMC St. Radboud, Nijmegen

REFERENCES:
- See also: Bladder Cancer Advocacy Network (BCAN) — http://www.bcan.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Ta/T1, Randomized to White Light Cystoscopy; Patients With Ta/T1 Randomized to Hexvix Cystoscopy: Patients with non-invasive papillary bladder cancer (Ta/T1), enrolled in the previously completed pivotal phase III study PCB305/04 who were followed for recurrence.
Period: Overall Study
Arm/Group | Patients With Ta/T1, Randomized to White Light Cystoscopy | Patients With Ta/T1 Randomized to Hexvix Cystoscopy
Started | 280 | 271
Completed | 261 | 255
Not Completed | 19 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With Ta/T1, Randomized to White Light Cystoscopy | Patients With Ta/T1 Randomized to Hexvix Cystoscopy | Total
Number analyzed (Participants) | 280 | 271 | 551
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (10.68) | 68 (10.79) | 68.8 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 59 | 116
  Male | 223 | 212 | 435

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Longer-term Recurrence-free Rates After Hexvix (Cysview) and Non-Hexvix (Cysview) Cystoscopy/TURB
Description: To extend the follow-up period of the pivotal trial (B305/04) to up in all available patients, to assess a longer-term estimate of recurrence-free rates after Hexvix and non-Hexvix cystoscopy/TURB, and to assess numbers and types of recurrences, amount and type of treatment given, and numbers of deaths.
Time Frame: up to 5.5 years retrospectively
Population: ITT
Measure: Number; unit: percentage of paticipants
Arm/Group | Patients With Ta/T1, Randomized to White Light Cystoscopy | Patients With Ta/T1 Randomized to Hexvix Cystoscopy
Number analyzed (Participants) | 261 | 255
percentage of paticipants | 38 | 31.8
Statistical Analysis 1: Comparison: Patients With Ta/T1, Randomized to White Light Cystoscopy; Test type: Superiority or Other; p = 0.141, Fisher Exact

2. Other Pre Specified Outcome: Median Time to Recurrence
Time Frame: up to 4.5 years
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Patients With Ta/T1, Randomized to White Light Cystoscopy | Patients With Ta/T1 Randomized to Hexvix Cystoscopy
Number analyzed (Participants) | 261 | 255
months | 9.4 [6.83 to 12.87] | 16.4 [11 to 25]
Statistical Analysis 1: Comparison: Patients With Ta/T1, Randomized to White Light Cystoscopy; Test type: Superiority or Other; p = 0.041, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Recurrence Free Survival
Time Frame: up to 4.5 years
Population: Intention-to-treat (ITT)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Patients With Ta/T1, Randomized to White Light Cystoscopy | Patients With Ta/T1 Randomized to Hexvix Cystoscopy
Number analyzed (Participants) | 261 | 255
months | 9.6 [7.00 to 13.33] | 16.4 [11.8 to 25.00]
Statistical Analysis 1: Comparison: Patients With Ta/T1, Randomized to White Light Cystoscopy; Test type: Superiority or Other; p = 0.056, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Rate of Progression
Description: Only patients with Ta/T1 were included in the follow-up study. "Progression" is defined as presence of T2-T4 tumors, with or without carcinoma in situ (CIS), at worst recurrence.
Time Frame: 4.5 years
Measure: Number; unit: percentage of patients
Arm/Group | Patients With Ta/T1, Randomized to White Light Cystoscopy | Patients With Ta/T1 Randomized to Hexvix Cystoscopy
Number analyzed (Participants) | 261 | 255
percentage of patients | 6.1 | 3.1

ADVERSE EVENTS:
Description: There was no treatment in this clinical study, only a follow-up of previously treated patients, so assessment of safety was not applicable.
Arm/Group | Patients With Ta/T1 Randomized to Hexvix Cystoscopy | Patients With Ta/T1, Randomized to White Light Cystoscopy
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days